CLINICAL TRIAL: NCT03422575
Title: Bioequivalence Study of 120 mg Etoricoxib Film-coated Tablet Produced by PT Dexa Medica in Comparison With the Comparator Drug (Arcoxia® Film-coated Tablet 120 mg, Frosst Iberica S.A., Spain, for Merck Sharp & Dohme (Australia) Pty Limited, Australia, Registered by PT Schering-Plough Indonesia, Tbk.)
Brief Title: Bioequivalence Study of 120 mg Etoricoxib Film-coated Tablets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Collaborators: PT Equilab International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 369/EQL/2015
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Healthy
MeSH Terms: interventions — Etoricoxib

STUDY DESIGN:
Intervention Model Description: This was a bioequivalence study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Etoricoxib 120Mg film-coated Tablet at single dose was given to subjects in this arm.
  Interventions: Drug: Etoricoxib 120Mg Film-coated Tablet
- Reference (Active Comparator): Arcoxia® 120 mg Film-coated tablet (Frosst Iberica S.A., Spain for Merck Sharp & Dohme (Australia) Pty Limited, Australia, registered by PT. Schering-Plough Indonesia Tbk) was given to subjects in this arm.
  Interventions: Drug: Arcoxia® 120 mg Film-coated tablet (Frosst Iberica S.A., Spain for Merck Sharp & Dohme (Australia) Pty Limited, Australia, registered by PT. Schering-Plough Indonesia Tbk)

INTERVENTIONS:
Drug: Etoricoxib 120Mg Film-coated Tablet — One tablet of the Test drug was given orally (swallowed with 200 mL of water, without chewing), after an overnight fast, and after fasting (pre-dose) blood-sampling.
  Other Names: Test
  Arms: Test
Drug: Arcoxia® 120 mg Film-coated tablet (Frosst Iberica S.A., Spain for Merck Sharp & Dohme (Australia) Pty Limited, Australia, registered by PT. Schering-Plough Indonesia Tbk) — One tablet of the Reference drug was given orally (swallowed with 200 mL of water, without chewing), after an overnight fast, and after fasting (pre-dose) blood-sampling.
  Other Names: Reference
  Arms: Reference

SUMMARY:
The present study was a randomized, open-label, two-period, two-sequence, cross-over study, conducted to find out whether the etoricoxib 120 mg film-coated tablet produced by PT Dexa Medica (test drug) was bioequivalent to the reference drug (Arcoxia® Film-Coated Tablet 120 mg, PT. Schering-Plough Indonesia Tbk), under fasting condition with a fourteen days wash-out period, involving 26 healthy adult male and female subjects.

DETAILED DESCRIPTION:
This was a randomized, open-label, two-period, two-sequence, cross-over study under fasting condition with a fourteen days wash-out period, involving 26 healthy adult male and female subjects. The participating subjects had an overnight fast and in the next morning were given orally either one film-coated tablet of the test drug or one film-coated tablet of the reference drug with 200 mL of water. Blood samples were drawn immediately before taking the drug (baseline), and at 15, 30, and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, and 72 hours after drug administration, analysed for plasma concentrations of etoricoxib and used to evaluate the pharmacokinetics parameters of the single dose administration. After a fourteen-day washout period, the procedure was repeated using the alternate drug. The plasma concentrations of etoricoxib were determined by using a high pressure liquid chromatography with ultraviolet detection (HPLC-UV) method.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects Healthy was defined as the absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening.
2. Aged 18 - 55 years inclusive.
3. Preferably non-smokers or smoke less than 10 cigarettes per day.
4. Able to participate and would provide written informed consent to participate.
5. BMI within 18 to 25 kg/m2.
6. Vital signs (after 10 minutes rest) were within the following ranges:

SBP 100 - 120 mmHg ; DBP 60 - 80 mmHg; HR 60 - 90 bpm.

Exclusion Criteria:

1. Personal/family history of allergy or hypersensitivity or contraindication to etoricoxib or allied drugs.
2. Pregnant or lactating women.
3. Any major illness in the past 90 days or clinically significant ongoing chronic illness
4. Presence of any clinically significant abnormal laboratory values during screening.
5. Positive Hepatitis B surface antigen (HBsAg), anti-HCV, or anti-HIV.
6. Clinically significant hematology abnormalities.
7. Clinically significant electrocardiogram (ECG) abnormalities.
8. Any surgical or medical condition (present or history) which might significantly alter the absorption, distribution, metabolism or excretion of the study drug, e.g. gastrointestinal disease including gastric or duodenal ulcers or history of gastric surgery.
9. Past history of anaphylaxis or angioedema.
10. History of drug or alcohol abuse within 12 months prior to screening for this study.
11. Participation in any clinical trial within the past 90 days calculated from the last visit.
12. History of any bleeding or coagulative disorders.
13. History of difficulty with donating blood or difficulty in accessibility of veins in left or right arm.
14. A donation or loss of 300 mL (or more) of blood within 3 months before this study's first dosing day.
15. Intake of any prescription, non-prescription drug, food supplement or herbal medicine within 14 days of this study's first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | 72 hours
  The area under plasma concentration-time curve from time zero to last observed concentration truncated at 72-hour (AUC0-72h)
Cmax | 72 hours
  Maximum plasma concentration

SECONDARY OUTCOMES:
Tmax | 72 hours
  Time to maximum plasma concentration
T1/2 | 72 hours
  The terminal half-life

CONTACTS AND LOCATIONS:
Overall Officials: Effi Setiawati, MSc, Study Director — Equilab International
Locations (1):
- PT Equilab International, Jakarta, Indonesia